CLINICAL TRIAL: NCT01488942
Title: A Randomized Clinical Trial Evaluating the Role of Contingent Reinforcement in the Engagement of and Retention of Drug Users in HAART Programs
Brief Title: Use of Incentives to Retain Drug Users in HIV Therapy
Acronym: Incentives-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark Hull, Clinical Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H11-00514; 1R01DA031043-01 (NIH); H11-00514 (Other: University of British Columbia)
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: HIV Infection
Keywords: HIV; reinforcement; medication adherence; patient compliance; antiretroviral therapy, highly active
MeSH Terms: conditions — HIV Infections; Medication Adherence; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- monetary reinforcer (Experimental): Subjects randomized to this arm will receive an escalating reinforcer initially for attendance at each clinic visit (until month 6 after starting HAART) and subsequently (until month 12 after starting HAART) will receive an escalating variable reinforcer for each month in which a viral load at or below 100 copies/mL is maintained
  Interventions: Other: monetary reinforcer
- no reinforcer (No Intervention): All subjects will receive HAART and standard medical care, but subjects in the control arm will not receive monetary reinforcers.

INTERVENTIONS:
Other: monetary reinforcer — The protocol will follow an escalating schedule of reinforcements tied to clinic visit attendance for the first 24 weeks, after which the reinforcers will take the form of an escalating variable reinforcement schedule in the form of fishbowl prize draws linked to maintenance of suppressed viral load for the remainder of the 52-week study period. In addition, a reset function will be incorporated by which the reinforcer will be rolled back to an initial lower value if clinic visits or viral load targets are not met. This will be rapidly scaled up again once targets are met.
  Other Names: contingency management
  Arms: monetary reinforcer

SUMMARY:
In many urban centres including Vancouver's Downtown Eastside, there is a high rate of HIV infection among users of illicit drugs. Among drug users who present to care and start highly active antiretroviral therapy (HAART), retention in care and adherence to their treatment regimen may be less than optimal. Given the known benefits of HAART on both the individual and populational levels, new strategies are required to help retain HIV-infected drug users on HAART.

Contingency management (CM) is a strategy to affect behaviour by providing a reward (e.g. money) to reinforce the desired behaviour. CM has been used with success in other areas of medicine (e.g. smoking cessation, weight loss) and in the drug using population, but has not been established as a means to improve retention in HAART programs.

The proposed research primarily seeks to assess the effectiveness of monetary-based CM in retaining HIV-infected drug users in HAART programs. 240 HAART-eligible subjects will be randomized in a 2:1 ratio to either receive (n=160) the reinforcer or to a control arm (n=80). All subjects will receive HAART and standard care, and those randomized to the reinforcer arm will receive escalating reinforcement initially for attendance at each clinic visit (until month 6 after starting HAART) and subsequently (until month 12 after starting HAART) will receive an escalating variable reinforcer for each month in which a plasma viral load less than or equal to 100 copies/mL is maintained.

Our hypotheses are that drug users initiating HAART and randomly selected to receive a reinforcer for attending clinic visits then maintaining monthly virologic suppression during the first 52 weeks after HAART initiation will be significantly more likely to achieve virologic suppression at 52 weeks, will have a significantly longer duration of sustained virologic suppression during the first 52 weeks, and will be significantly more likely to maintain virologic suppression at 72 weeks after HAART initiation, than those not offered a reinforcer.

DETAILED DESCRIPTION:
Once HAART has been initiated, participants will be expected to be assessed at weeks 1,2,3,4,6,8,10,12,14, and 16. Detailed adherence and dispensing records for all antiretroviral medications for each participant will be maintained. Adherence will be assessed primarily on the basis of pharmacy refill records, as well as self-report. Subsequently participants will attend monthly clinical follow-up visits at weeks 20, 24, 28, 32, 36, 40, 44, 48, and 52. Standard laboratory monitoring will be performed at that time, and will include complete blood count (CBC), differential, basic chemistry, liver and kidney profile, as well as CD4 cell count and plasma HIV-1-RNA level, consistent with current care guidelines. All patients will also undergo urine toxicology screens at baseline and quarterly (weeks 12, 24, 36, and 52) in order to assess any effects of engaging in HAART programs on substance use. Follow-up will also include an adverse events assessment (ADE) from a standardized list of signs and symptoms noted by either the patient or practitioner or identified through laboratory testing. At baseline and each quarterly visit, participants will complete the Center for Epidemiologic Studies Depression Scale (CES-D) where a score of 16 correlates with risk of depression. This tool has been validated in our population in a prior study. Participants will also complete the Addiction Severity Index questionnaire, a validated instrument used to examine severity of psychosocial problems in seven domains including drug and alcohol use . Composite scores are derived, and higher scores reflect greater problems. Past 3-month versions of the HIV Risk Behavior Scale will also be administered at baseline and at quarterly visits. This scale assesses injection drug use and sexual behaviors, and responses are coded on a 6-point scale with higher values indicating higher risk.

Participants who are randomized to receive a reinforcer for clinic follow-up will receive the reinforcer at the end of each clinic visit. When the reinforcer is linked to plasma viral load, subjects in the reinforcer arm will be notified within a week of the plasma viral load result, and of any reinforcement earned. Subjects can elect to come in at any time to receive the reinforcement, or they can wait until their next monthly appointment and receive the earnings at that time.

For participants who do not present for laboratory and clinical follow-up within two weeks on either side of their scheduled quarterly visit, an extensive investigation into the client's whereabouts through street outreach as well as a search of hospital records for hospitalization and the provincial vital statistics database for possible deaths will be prompted. Those who discontinue therapy or who are lost to follow-up at or before 52 weeks will be considered therapy failures in the analyses.

A final visit 24 weeks after the week 52 visit will be performed. This will involve the same procedures as the quarterly study visits during the first year, including standard laboratory tests and urine toxicology, ADE assessments, and CES-D, Addiction Severity Index and HIV Risk Behavior Scale questionnaires. Participants who fail to present for laboratory and clinical follow-up within 2 weeks of the expected date of this visit will be sought as described above.

ELIGIBILITY:
Inclusion Criteria:

1. Adults at least 19 years of age.
2. Have used illicit drugs (heroin, cocaine, cocaine/heroin combinations, methamphetamines, injectable morphine and codeine, but excluding isolated marijuana use) at least once in the past three months.
3. Eligible for, and willing to initiate HAART. To be eligible for HAART, participants must have CD4 count at or below 350 cells/mm3 at the HAART eligibility screening visit and/or significant co-morbidities identified in current international guidelines (hepatitis B/C co-infection, HIV associated nephropathy, high risk for cardiovascular disease)

Exclusion Criteria:

1. No history of active drug use as defined above.
2. Pregnant women.
3. Receipt of HAART for more than 6 months within the preceding 12 months.
4. Persons in recovery from gambling addiction (due to the element of chance in the CM intervention).
5. Persons acutely intoxicated at time of consent.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2012-12; Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
proportion of subjects achieving virologic suppression (plasma viral load less than or equal to 100 copies/mL) at 52 weeks after HAART initiation. | 52 weeks after HAART initiation.

SECONDARY OUTCOMES:
duration of sustained virologic suppression during the first 52 weeks after HAART initiation. | during the first 52 weeks after HAART initiation.
  Virologic response will be defined as the percentage of follow-up time with plasma viral load less than or equal to 100 copies/mL.
proportion of subjects achieving virologic suppression (plasma viral load less than or equal to 100 copies/mL) at 72 weeks after HAART initiation. | 72 weeks after HAART initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hull, MD, Principal Investigator — University of British Columbia; Julio SG Montaner, MD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, VIDUS and Incentives study office site, 611 Powell St., Vancouver, British Columbia, Canada